CLINICAL TRIAL: NCT05696561
Title: A Prospective, Multicenter, First in Human Clinical Trial to Evaluate the Safety and Effectiveness of the DF12 CANALOPLASTY AND TRABECULOTOMY SURGICAL SYSTEM in Subjects With Open-Angle Glaucoma Undergoing Cataract Surgery
Brief Title: Clinical Trial to Evaluate the Safety and Effectiveness of a Canaloplasty Device in Subjects With Open-Angle Glaucoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New World Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DF12-CL-22-01
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-04

CONDITIONS: POAG

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment with a Canaloplasty Device (Experimental): Canaloplasty Device
  Interventions: Device: Canaloplasty Device

INTERVENTIONS:
Device: Canaloplasty Device — Canaloplasty

SUMMARY:
Clinical Trial to Evaluate the Safety and Effectiveness of a Canaloplasty Device in Subjects with Open-Angle Glaucoma

ELIGIBILITY:
Inclusion Criteria:

1. Subjects qualifying for cataract surgery
2. Subjects with diagnosis of open-angle glaucoma in at least one eye with unmedicated IOP of 22-34 mmHg.

Exclusion Criteria:

1. Patients who cannot be washed-out of IOP-lowering medications.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
IOP change | Month6
  proportion of treated eyes with > 20% change in unmedicated IOP

SECONDARY OUTCOMES:
IOP | Months 6 and 12
  Change in IOP
IOP meds | Month 6 and 12
  Change in number of IOP lowering medications

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sun, PhD, Study Director — New World Medical, Inc.
Locations (3):
- Clinica 20/20, San José, Costa Rica
- Centro Oftalmologico Robles, Santa Rosa de Copán, Honduras
- Laser y Ultrasonido Ocular, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No